CLINICAL TRIAL: NCT06464549
Title: Spontaneous Eye Blinking Evaluation for Cognitive Assessment of Individuals With Severe Acquired Brain Injury
Acronym: SEE-ABI
Status: Active, not recruiting | Type: Observational
Sponsor: Alfonso Magliacano (Other)
Responsible Party: Sponsor-Investigator, Alfonso Magliacano, Researcher, Fondazione Don Carlo Gnocchi Onlus
Organization: Fondazione Don Carlo Gnocchi Onlus (Other)
Other Study IDs: SEE-ABI
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Disorders of Consciousness; Acquired Brain Injury
Keywords: severe acquired brain injury; cognitive rehabilitation; diagnosis; eye blinking; machine learning
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with severe acquired brain injury: Patients' inclusion criteria: (i) age≥18 years; (ii) time post-injury≥28 days. Exclusion criteria will be: (i) large craniectomy interfering with EEG recording; (ii) unstable clinical conditions; (iii) presence of ophthalmic disorders, or central or peripheral impairments in eyelid motility on clinical evaluation; (iv) administration of sedative medication in the previous 24h; (v) previous history of neurological or psychiatric diseases; (vi) written informed consent by patient or, where necessary, by primary caregiver.
  Interventions: Diagnostic Test: EEG-EOG recording at rest and during an auditory oddball paradigm
- Benchmark sample: i) age≥18 years; ii) normal or corrected-to-normal vision excluding contact lenses; iii) a total score >22.23 at the Montreal Cognitive Assessment (Santangelo et al., 2015); iv) written informed consent. Exclusion criteria: i) presence of ophthalmic disorders, or central or peripheral impairments in eyelid motility on clinical evaluation; ii) consumption of drugs acting on the central nervous system; iii) previous history of neurologic or psychiatric diseases.
  Interventions: Diagnostic Test: EEG-EOG recording at rest and during an auditory oddball paradigm

INTERVENTIONS:
Diagnostic Test: EEG-EOG recording at rest and during an auditory oddball paradigm — Participants will attend an electroencephalogram-electrooculogram (EEG-EOG) recording session. Eye blinking will be examined during a rest condition (duration: 8 min) and during an active auditory oddball task (duration: 8 min), consisting of randomly intermixed tones (non-target: 500 Hz, overall probability: 80%, n=312; target: 1000 Hz, overall probability: 20%, n=78) presented with a 1-s inter-stimulus interval through headphones.

SUMMARY:
Assessment of consciousness and attention in individuals with severe Acquired Brain Injury (sABI) is crucial for planning rehabilitation, but it is often hindered by coexisting sensory-motor and/or cognitive-behavioural disorders.

This project aims at evaluating the value of spontaneous eye blinking features to assess patients' attentional abilities and to distinguish patients with unresponsive wakefulness syndrome (UWS) from those in minimally conscious state (MCS).

Patients will undergo an EEG-EOG recording at rest and during an auditory oddball task. Eye blinking features on EOG will be analysed and compared to that of healthy individuals. A machine-learning-based algorithm using blinking features for the diagnosis of patients with sABI will be studied and validated preliminarily.

This project will help to stratify patients with sABI using easy-to-detect clinical markers, supporting clinicians' decision-making about patient's management. Additionally, blinking patterns related to residual attentional abilities in patients emerged from disorders of consciousness will be investigated.

DETAILED DESCRIPTION:
Overall aim: to provide preliminary results on the value of spontaneous eye blinking features (i.e., rate, amplitude, duration, and variability in intervals between blinks), which do not rely on voluntary behavioural responses, for improving the assessment of attentional abilities and consciousness in patients with sABI.

Specific aims:

1. to confirm the diagnostic value of EBR in pDoC patients, as in Magliacano et al.'s (2021) study;
2. to improve diagnostic accuracy of patients with prolonged Disorders of Consciousness (pDoC) by evaluating additional blinking features (i.e., amplitude, duration, variability in intervals between blinks) for discriminating patients in UWS from those in MCS or conscious.
3. to explore the usefulness of eye blinking features analysis for assessing residual attentional abilities in full-conscious patients recovering from pDoC.
4. prototyping a machine-learning-enabled pipeline for supporting consciousness diagnosis based on Eye Blink Rate (EBR) and EOG-derived features. The interpretability and reliability aspects will be carefully evaluated to obtain a clinically usable solution for supporting diagnostic procedures and planning tailored cognitive rehabilitation.

Overall, this study is proposing a preliminary investigation, with pilot samples of both healthy and test population, for the analysis of EBR and EOG-derived biomarkers. These results will lay the foundations for the development and validation of multifactorial decisional algorithms for patients' diagnostic and prognostic stratification, based on easily collectable clinical markers.

This project has an observational, cross-sectional design. All patients with sABI consecutively admitted will be screened. We plan to enrol a convenience test sample of 35 patients with sABI including 10 patients with pDoC (5 in UWS, 5 in MCS) and 25 patients who recovered full consciousness after sABI.

A benchmark population of 20 healthy individuals, balanced for age and sex with the patient sample, will be also enrolled, by means of word-of-mouth according to a snowball sampling. This population will undergo anamnestic interview, and neurological and primary cognitive examination for excluding history or presence of neurological disorders. At study entry, patients' demographic (e.g., age, sex), anamnestic (e.g., aetiology, time post-injury, brain lesion location), and clinical data will be collected. Patients' clinical diagnosis and cognitive functioning will be classified according to their best score on the repeated Coma Recovery Scale-Revised (CRS-R) and on Levels of Cognitive Functioning (LCF), respectively.

Within 2 weeks from study entry, each patient will attend an electroencephalogram-electrooculogram (EEG-EOG) recording session. Eye blinking will be examined during a rest condition (duration: 8 min) and during an active auditory oddball task (duration: 8 min), consisting of randomly intermixed tones (non-target: 500 Hz, overall probability: 80%, n=312; target: 1000 Hz, overall probability: 20%, n=78) presented with a 1-s inter-stimulus interval through headphones. To complement clinical assessment, the background activity on resting EEG and the presence of the P300 component on event-related potentials following the auditory oddball paradigm will be evaluated. Patients' consciousness (CRS-R) and cognitive functioning (LCF) levels will be gathered on the day of the EEG-EOG recording session, and considered for statistical analysis.

Control participants will undergo the same EEG-EOG recording as the patients. For both participant groups, blinks will be defined as a sharp positive peak followed by a shallow negative deflection in a time window of <400 ms on the EOG. Moreover, to prevent awareness of blink recording affects blink features, throughout recording sessions participants will be never informed of the blinking recording, but they will be encouraged to stay relaxed with their eyes open. This procedure will be conducted regardless of the participant (patient or control) group.

Biostatistical analyses will be exploited for the investigation of associations between EOG-derived biomarkers and residual attentional abilities in conscious sABI patients under different acquisition paradigms, in response to Objective 3. Objective 4 will be addressed through the development of Machine Learning-based prototypes for the diagnosis of patients with pDoC using information derived from EOG signals, complemented by EEG and clinical data. The interpretability and error analyses will pose the premises for the identification of eventual covert patterns contained in EOG data.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of severe acquired brain injury;
* age≥18 years;
* time post-injury≥28 days
* written informed consent by patient or, where necessary, by primary caregiver

Exclusion criteria will be:

* large craniectomy interfering with EEG recording;
* unstable clinical conditions;
* presence of ophthalmic disorders, or central or peripheral impairments in eyelid motility on clinical evaluation;
* administration of sedative medication in the previous 24h;
* previous history of neurological or psychiatric diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with sABI consecutively admitted will be screened.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised | Within 2 weeks from study entry
  The Coma Recovery Scale-Revised is a clinical scale with a total score ranging from 0 to 23, with higher scores indicating a higher level of consciousness
Levels of Cognitive Functioning | Within 2 weeks from study entry
  Levels of Cognitive Functioning is a clinical scale with a score ranging from 1 to 8, with higher scores indicating a higher level of cognitive functioning

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Polo Specialistico Riabilitativo Fondazione Don Carlo Gnocchi ONLUS, Sant'Angelo dei Lombardi, AV
  - IRCCS Fondazione Don Carlo Gnocchi Firenze, Florence

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Magliacano A, Rosenfelder M, Hieber N, Bender A, Estraneo A, Trojano L. Spontaneous eye blinking as a diagnostic marker in prolonged disorders of consciousness. Sci Rep. 2021 Nov 17;11(1):22393. doi: 10.1038/s41598-021-01858-3. PMID 34789832